CLINICAL TRIAL: NCT02555787
Title: Global Multicentre Kidney Transplant Advagraf Conversion Registry. A Non-interventional Post-authorisation Study (PAS)
Brief Title: Global, Multicentre, Non Interventional Advagraf Conversion Registry in Kidney Transplant Patients
Acronym: CHORUS
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 506-MA-1002
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation
Keywords: FK506E; Tacrolimus; Observational; Kidney transplantation; Advagraf
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients converted from tacrolimus BD to Advagraf: Oral
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: FK506E; Advagraf; Astagraf XL; Prograf XL

SUMMARY:
A study to evaluate changes over time in renal function from baseline (time of conversion) up until five years post conversion in kidney transplant patients converted from tacrolimus twice daily (BD) formulations to a once daily formulation as Advagraf.

DETAILED DESCRIPTION:
This is a multicenter long-term (up to five years post-conversion), non-interventional registry in kidney transplant patients who have been converted from tacrolimus BD to Advagraf. Centers that are providing medical care for kidney transplant patients who may convert patients from tacrolimus BD to Advagraf will be identified and requested to approach patients for consent to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant patients who are on tacrolimus BD and identified for conversion to Advagraf. Patients will only be approached about participating in the registry after their physician has made the decision to convert them to Advagraf. Patients previously treated with Advagraf and who have stopped for any reason will not be excluded from the registry provided that the physician has decided to convert.

Exclusion Criteria:

* Patients currently taking Advagraf treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Probability Sample
Enrollment: 4430 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in renal function as measured by eGFR using the MDRD-4 formula | At transplantation, within 3 months after transplantation, up to 2 years pre-conversion and then every 6 months prior to conversion, at conversion (baseline), 12 months post-conversion and annually thereafter until EOS (up to 5 years post conversion)
  Estimated Glomerular Filtration Rate (eGFR), Modification Diet in Renal Disease (MDRD-4), End of Study (EOS)

SECONDARY OUTCOMES:
Change in renal function as measured by eGFR using the CKD-Epi formula | At transplantation, within 3 months after transplantation, up to 2 years pre-conversion and then every 6 months prior to conversion, at conversion (baseline), 12 months post-conversion and annually thereafter until EOS (up to 5 years post conversion)
  Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi)
Overall patient survival | From transplantation to EOS (up to 5 years post conversion) or date of death from any cause
  Patients who are lost to follow up or alive at EOS - or at time of analysis will be censored
Overall graft survival (time to graft loss) | From transplantation to date of graft loss
  Defined as time from transplantation to graft loss. Graft loss is defined as re-transplantation, nephrectomy, death or as dialysis ongoing at end of study or at the time of discontinuation of the patient from the study. The date of graft loss is the earliest date of any of these events. In case of dialysis as reason for graft loss, the date of graft loss is the first day of the last ongoing dialysis period reported
DSA status (de novo) | From transplantation to EOS (up to 5 years post conversion)
  Donor Specific Antibody (DSA). Laboratory assessment performed where possible in accordance with standard of care
Incidence of BPAR episodes | From transplantation to EOS (up to 5 years post conversion)
  Biopsy Proven Acute Rejection (BPAR). Severity by Banff classification (International standardisation of criteria for histological diagnosis of allograft rejection), treated and untreated, and steroid sensitive or resistant
Time to first incidence of BPAR episodes | From transplantation to EOS (up to 5 years post conversion)
  Severity by Banff classification, treated and untreated, and steroid sensitive or resistant
Advagraf dose | From transplantation to EOS (up to 5 years post conversion)
Tacrolimus trough level | From transplantation to EOS (up to 5 years post conversion)
Current immunosuppressant regimen | From transplantation to EOS (up to 5 years post conversion)
  Dose and formulation (additional to or instead of Advagraf)
Status of treatment with Advagraf | From transplantation to EOS (up to 5 years post conversion)
  Patients who discontinued Advagraf treatment will be retained in the registry for data on long-term outcomes provided consent is not withdrawn. The reasons associated with the discontinuation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs Europe, Study Director — Astellas Pharma Europe Ltd.
Locations (129):
- Australia (8):
  - Site AU6107, Camperdown, New South Wales
  - Site AU6106, Gosford, New South Wales
  - Site AU6104, New Lambton, New South Wales
  - Site AU6103, Westmead, New South Wales
  - Site AU6111, Harvey Bay, Queensland
  - Site AU6108, North Adelaide, South Australia
  - Site AU6110, Nedlands, Western Australia
  - Site AU6105, Perth, Western Australia
- Austria (4):
  - Site AT4301, Graz, Styria
  - Site AT4302, Innsbruck, Tyrol
  - Site AT4303, Innsbruck, Tyrol
  - Site AT4304, Linz, Upper Austria
- Site BE3201, Leuven, Vlaams Brabant, Belgium
- Site CA1001, Vancouver, British Columbia, Canada
- Site CZ4202, Olomouc, Czechia
- France (23):
  - Site FR3310, Nice, Alpes-Maritimes
  - Site FR3318, Strasbourg, Alsace
  - Site FR3324, Lyon, Auvergne-Rhône-Alpes
  - Site FR3315, Marseille, Bouches-du-Rhône
  - Site FR3303, Caen, Calvados
  - Site FR3306, Besançon, Doubs
  - Site FR3311, Brest, Finistère
  - Site FR3302, Bordeaux, Gironde
  - Site FR3313, Toulouse, Haute-Garonne
  - Site FR3307, Rouen, Haute-Normandie
  - Site FR3321, Limoges, Hautte-Vienne
  - Site FR3317, Rennes, Ille-et-Vilaine
  - Site FR3305, Tours, Indre-et-Loire
  - Site FR3312, Nantes, Loire-Atlantique
  - Site FR3314, Angers, Maine-et-Loire
  - Site FR3325, Lille, Nord
  - Site FR3309, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Site FR3308, Amiens, Picardie
  - Site FR3319, Clermont-Ferrand, Puy-de-Dôme
  - Site FR3322, Poitiers, Vienne
  - Site FR3323, Paris
  - Site FR3301, Créteil, Île-de-France Region
  - Site FR3316, Le Kremlin-Bicêtre, Île-de-France Region
- Germany (3):
  - Site DE4902, Mannheim, Baden-Wurttemberg
  - Site DE4901, Würzburg, Bavaria
  - Site DE4903, Hanover, Lower Saxony
- Greece (2):
  - Site GR3002, Athens
  - Site GR3004, Athens
- Hong Kong (2):
  - Site HK8201, Hong Kong
  - Site HK8521, Hong Kong
- Hungary (2):
  - Site HU3601, Debrecen, Hajdú-Bihar
  - Site HU3602, Budapest
- Italy (17):
  - Site IT3903, Napoli, Campania
  - Site IT3907, Verona, Veneto
  - Site IT3905, Bari
  - Site IT3902, Bologna
  - Site IT3914, Bolzano
  - Site IT3901, Genova
  - Site IT3904, L’Aquila
  - Site IT3911, Novara
  - Site IT3916, Novara
  - Site IT3910, Padua
  - Site IT3909, Perugia
  - Site IT3912, Salerno
  - Site IT39013, Salerno
  - Site IT3913, Salerno
  - Site IT3908, Sassari
  - Site IT3915, Udine
  - Site IT3906, Venezia
- Japan (10):
  - Site JP8108, Nagoya, Aiti
  - Site JP8109, Toyoake, Aiti
  - Site JP8107, Chiba, Chiba
  - Site JP8110, Nishinomiya, Hyôgo
  - Site JP8111, Nishinomiya, Hyôgo
  - Site JP8106, Kawasaki-shi, Kanagawa
  - Site JP8105, Ōta-ku, Tôkyô
  - Site JP8104, Shinjuku-Ku, Tôkyô
  - Site JP8101, Akita
  - Site JP8102, Niigata
- Site MY6001, Kuala Lumpur, Wilayah Persekutuan Kuala Lump, Malaysia
- Netherlands (4):
  - Site NL3103, Nijmegen, Gelderland
  - Site NL3104, Amsterdam, North Holland
  - Site NL3105, Groningen
  - Site NL3101, Utrecht
- Site PH6303, Quezon City, National Capital Region, Philippines
- Poland (4):
  - Site PL4806, Poznan, Greater Poland Voivodeship
  - Site PL4808, Lublin, Lublin Voivodeship
  - Site PL4801, Warsaw, Masovian Voivodeship
  - Site PL4807, Szczecin, West Pomeranian Voivodeship
- Site PT3511, Porto, Portugal
- Romania (4):
  - Site RO4004, Cluj-Napoca, Cluj
  - Site RO4001, Bucharest
  - Site RO4002, Bucharest
  - Site RO4003, Bucharest
- Serbia (4):
  - Site SB3804, Niš, Nišavski Okrug
  - Site SB3801, Belgrade
  - Site SB3802, Belgrade
  - Site SB3803, Novi Sad
- South Korea (18):
  - Site KR8214, Busan, Busan Gwang'yeogsi [Pusan-Kwan
  - Site KR8205, Busan, Busan Gwang'yeogsi [Pusan-Kwan
  - Site KR8203, Pusan, Busan Gwang'yeogsi [Pusan-Kwan
  - Site KR8202, Daegu, Daegu Gwang'yeogsi [Taegu-Kwan
  - Site KR8219, Daegu, Daegu Gwang'yeogsi
  - Site KR8207, Daejeon, Daejeon Gwang'yeogsi [Taejon-K
  - Site KR8212, Gwangju, Gwangju Gwang'yeogsi
  - Site KR8218, Suwon, Gyeonggido [Kyonggi-do]
  - Site KR8216, Bucheon-si, Gyeonggido
  - Site KR8201, Incheon, Incheon Gwang'yeogsi [Inch'n-K
  - Site KR8211, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Site KR8210, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Site KR8206, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Site KR8209, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Site KR8204, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Site KR8208, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Site KR8213, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Site KR8215, Ulsan, Ulsan Gwang'yeogsi [Ulsan-Kwan
- Spain (3):
  - Site ES3410, Santiago de Compostela, A Coruña
  - Site ES3401, Barcelona
  - Site ES3403, Barcelona
- Taiwan (3):
  - Site TW8862, Kaohsiung City, Kaohsiung
  - Site TW8863, Taichung, Taichung Municipality
  - Site TW8861, Tainan
- Thailand (3):
  - Site TH6601, Bangkok, Krung Thep Maha Nakhon [Bangko
  - Site TH6602, Bangkok, Krung Thep Maha Nakhon [Bangko
  - Site TH6603, Khon Kaen
- United Kingdom (7):
  - Site GB4403, Peterborough, Cambridgeshire
  - Site GB4405, Exeter, Devon
  - Site GB4406, Manchester, Lancashire
  - Site GB4407, Ipswich, Suffolk
  - Site GB4401, Leeds
  - Site GB4402, Liverpool
  - Site GB4408, London
- Vietnam (2):
  - Site VN8401, Hà Nội, Ha Noi, Thanh Pho
  - Site VN8402, Ho Chi Minh City, Ho Chi Minh, Thanh Pho

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.